CLINICAL TRIAL: NCT04857151
Title: Stress, Inflammation and Immune Response Pilot Study- Aim 3
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-1173- Aim 3; PRJ66UV (Other Grant/Funding Number: UNIVERSITY OF WISCONSIN FOUNDATION); A536300 (Other: UW Madison); SMPH/PATHOL & LAB MED (Other: UW Madison); Protocol version 08/29/2023 (Other: UW Madison)
Record Dates: First submitted 2021-04-08; First posted 2021-04-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus; Inflammation
Keywords: Neutrophil; Meditation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Control
- App based mindfulness program (ABMP) (Experimental): Participants in this group will participate in App based mindfulness program (ABMP)
  Interventions: Behavioral: App based mindfulness program (ABMP)

INTERVENTIONS:
Behavioral: App based mindfulness program (ABMP) — App based mindfulness program (ABMP)
  Arms: App based mindfulness program (ABMP)

SUMMARY:
The overall goal of this study is to investigate the effects of stress and glucose intake at the molecular level including gene expression, protein and functional analysis of immune cells in real time.

Aim 1- Characterizing the immune response after acute stress and glucose consumption Aim 2- Temporal mapping of the modulation of immune cell function via meditation Aim 3-Influence of meditative practice on lupus patients Aim 4-Influence of meditative practice on healthy subjects

Current Clinicaltrials.gov record, will be focused on Aim-3 only. Aim-3 will test whether meditation alters neutrophil function and inflammation in patients with lupus. Study team will investigate whether patient neutrophils have altered NET formation, phagocytosis, ROS signaling and migration after ABMP. Innate immune function via analysis of monocytes by flow cytometry will also be analyzed. Other immune cell responses including CD8 T cells will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Lupus diagnosis according to >4 ACR 1987 criteria or >4 SLICC 2012 criteria or a diagnosis confirmed by a board-certified rheumatologist
* Capacity to provide informed consent and ability to speak and read English
* BMI under 35
* Must have access to an iOS or android smartphone to allow daily use of an app

Exclusion Criteria:

* Currently participating in another clinical trial with intervention. Participation in observational clinical trials is not grounds for exclusion.
* History of significant systemic disease (eg. cancer, infection, hematological, renal, hepatic, coronary artery disease or other cardiovascular disease, endocrinological (diabetes), neurologic, rheumatologic, or gastrointestinal disease)
* Acute illness or evidence of clinically significant active infection
* Pregnant, breast feeding or less than 6 months post-partum
* Taking prescribed psychotropic or central nervous system altering medications
* History of a diagnosed Bipolar Disorder, Schizophrenia, or Schizoaffective Disorder, epilepsy or seizures
* Individuals who are currently undergoing a depressive episode. Can include those who are under treatment and not depressed currently.
* Excluded based upon the screening visit
* Use of nicotine
* Significant previous training or significant current practice in meditation
* Completed Mindfulness Based Stress Reduction (MBSR) in the past
* Current meditation practice. Judgment: Participants will be included or excluded at the PIs discretion due to wide variation in responses (e.g. 2 people answer yes, one practices mindfulness 2x/week for 2 years (exclude), the other attends regular religious services (include))
* Significant daily practice with other mind-body techniques
* Daily Yoga or Tai Chi Practice - exclude
* Other daily practice - judgment

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Lupus is about nine times more common in females than in males.
Enrollment: 3 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in neutrophil function as assessed by Neutrophil extracellular trap(NET) formation | Baseline and 8 weeks
Change in phagocytic index of neutrophils | Baseline and 8 weeks
  Neutrophil phagocytosis is measured by quantifying the ingestion of fluorescent zymosan or E.coli bioparticles using fluorescence microscopy. A phagocytic index is calculated to report the number of particles phagocytosed per cell.
Change in neutrophil function as assessed by reactive oxygen species (ROS) production | Baseline and 8 weeks
Change in neutrophils' migratory ability as assessed by change in neutrophils' velocity | Baseline and 8 weeks
  Neutrophil migration is assessed using time lapse microscopy. The migration patterns of individual neutrophils are measured using NIH Image J FIJI and velocity (μm/min) is measured.
Change in neutrophils' migratory ability as assessed by change in "distance travelled" by neutrophils | Baseline and 8 weeks
  Neutrophil migration is assessed using time lapse microscopy. The migration patterns of individual neutrophils are measured using NIH Image J FIJI and distance (μm) is quantified.
Change in the expression of stress-induced genes | Baseline and 8 weeks

SECONDARY OUTCOMES:
Change in inflammatory cytokines level | Baseline and 8 weeks
  Peripheral blood mononuclear cells (PBMC) and sub-populations including CD8 T cells and NK cells will be isolated from blood to study inflammatory cytokines level.
Change in expression of 'immune cells activation markers' | Baseline and 8 weeks
Change in the monocyte activation level | Baseline and 8 weeks
  Monocytes will be analyzed by flow cytometry for activation markers and other markers of cell function.
Change in the methylation pattern of stress-induced genes | Baseline and 8 weeks
Change in the gene expression pattern of stress induced genes | Baseline and 8 weeks
Change in the cytokine secretion level from immune cells | Baseline and 8 weeks

OTHER OUTCOMES:
Change in PROMIS-GH (Patient-Reported Outcomes Measurement Information System Global Health) score | Baseline and 8 weeks
  PROMIS self-report measures are intended to be completed by the respondent without help from anyone else.
  The PROMIS GH is comprised of 10 global items. Each item represents a different domain of health. Mental health and physical health summary scores are computed and standardized to the general population. Both these component scores and individual global items can be used to assess patients' perceptions of their health.
  PROMIS global health can be converted to raw scores between 4-20 that can be converted to a t-score of 16.2-67.7. A higher score reflects better functioning.
Change in State Trait Anxiety Inventory (STAI) Score | Baseline and 8 weeks
  The State Trail Anxiety Inventory is a 20 item questionnaire about how the participant is feeling. The total possible range of scores is 20-80 lower scores indicate less anxiety.
Change in Five Facet Mindfulness Questionnaire (FFMQ) | Baseline and 8 weeks
  FFMQ is a 39-item questionnaire scored on a 5 pt likert scale for a total possible range of scores 39-195 where higher scores indicate increased mindfulness.
Change in the Perceived Stress Scale | Baseline and 8 weeks
  The Perceived Stress Scale is a 10-item survey scored on a 5-pt likert scale for a total possible range of scores 0-40 where higher scores indicate increased perceived stress.
Change in PROMIS-Positive Affect Score | Baseline and 8 weeks
  The PROMIS-Positive Affect Score is based on a 15-item survey, each item scored on a 5-pt likert scale for a total possible range of scores 15-75 where higher score indicated higher positivity.
Change in PROMIS-Depression Score | Baseline and 8 weeks
  The PROMIS-Depression Score is based on a 6-item survey, each item scored on a 5-pt likert scale for a total possible range of scores 6-30 where higher score indicate increased depression.

CONTACTS AND LOCATIONS:
Overall Officials: David Beebe, PhD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No